CLINICAL TRIAL: NCT02078037
Title: Systemic Normothermia in Intracerebral Hemorrhage (ICH)
Acronym: SNICH
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-1407
Record Dates: First submitted 2014-02-21; First posted 2014-03-05 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral hemorrhage; Perihematomal edema; hemorrhage; normothermia
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arctic Sun cooling device (Experimental): The Arctic Sun device pads will be placed on the patient as per manufacturer's instructions. Patients, who cannot tolerate placement of all the pads for any given reason, will still be included in the study if they can maintain normothermia (normal body temperature). The total normothermia time for the study is five days. After 5 days, the attending physician will make clinical decisions based on the patient needs.The temperature goal for this study is 36.5 degree Celsius, but normothermia for the purpose of this study will be defined as a temperature of 35.5 - 37.5 degree Celsius. A thermometer mounted urinary catheter will be used for temperature monitoring and feedback to the Arctic Sun.
  Interventions: Device: Arctic Sun cooling device
- Standard of Care (Active Comparator): Patient will be given standard fever management (acetaminophen + cooling blanket at the discretion of the treating physician) initiated at a temperature of 38.5 degrees Celsius
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Arctic Sun cooling device — The Arctic Sun® 5000 Temperature management systems (Bard Medical), a non- invasive, surface cooling technology that allows rapid and precise manipulation of core body temperature will be employed to maintain normothermia (normal temperature) in patients with ICH randomized to the treatment group.
  Other Names: The Arctic Sun® 5000 Temperature management systems
  Arms: Arctic Sun cooling device
Other: Standard of Care — Patient will be given standard fever management (acetaminophen + cooling blanket at the discretion of the treating physician)
  Arms: Standard of Care

SUMMARY:
Patients with a supratentorial intracerebral hemorrhage will be randomly assigned to either the experimental group which will keep them at a normal body temperature or the standard of care group. The investigators propose to test the hypothesis that prophylactic forced normothermia in patients with ICH leads to less systemic inflammation and decreased perihematomal edema.

DETAILED DESCRIPTION:
This is a randomized device efficacy trial. Patients with a supratentorial intracerebral hemorrhage (ICH) admitted to the Cleveland Clinic Neurointensive Care Unit within 1 day of symptom onset and who have not experienced episodes of temperature elevation will be enrolled after consent. Patients randomized to the experimental arm, will have Artic Sun cooling pads applied to the torso and thighs for five days. The Arctic Sun device will keep the body temperature at the normal range of 35.5 - 37.5 degrees Celsius. Patients randomized to the active comparator arm will receive a standard of care treatment at the discretion of the treating physician. Patients will have hourly measurement of blood pressure, heart rate, respiratory rate, urine output, temperature (from the urinary catheter) shivering scale, and nursing neurological assessment. Glasgow coma scale, NIH Stroke Scale Score (NIHSS), telemetry monitoring and labs will also be performed daily. The investigators will also collect demographic information about the patients (i.e. age, gender, medical risk factors) and information regarding their current disease process.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with spontaneous supratentorial ICH >20 cc
2. Age 18 to 85 years of age
3. Consent from the patient or surrogate decision maker
4. Within 24 hours of onset of ictus

Exclusion Criteria:

1. Hemorrhage secondary to trauma, Arterio-venous malformation (AVM), aneurysm or Arterio-venous dural fistula
2. Moribund state and deemed unlikely to survive until study completion (5 days)
3. Patients with a don-not-resuscitate (DNR) order
4. Known infection at the time of admission (elevated white blood cell count (WBC) with identified infection source).
5. Evidence of a blood dyscrasia
6. Pregnancy
7. Renal failure (CCR < 50 ml/min)
8. Contraindications for a brain MRI scan
9. Infratentorial ICH
10. Warfarin-induced intracerebral hemorrhages NOT corrected to International Normalized Ratio (INR) < 1.4 within 24 hours
11. Episode of fever > 38.5 degrees Celsius prior to enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
MRI measurement of relative perihematomal edema (% change of perihematomal edema) | First 5 days of hospital course
  Percent relative perihematomal edema growth between the initial MRI and the 5 day MRI

SECONDARY OUTCOMES:
Structured telephone interview of functional and cognitive outcome | 3 months and 1 year
  Functional and cognitive outcomes measured by structured phone assessment.
Serum cytokine measurement with inflammatory cytokine protein array | 5 days
  Cytokine markers of inflammation tested daily over the first 5 days.

OTHER OUTCOMES:
Serum cytokine measurement with inflammatory cytokine protein array in control ICH patients | 5 days
  Cytokine markers of inflammation tested daily over the first five days of the study in control ICH patients to determine the natural inflammation history of ICH.
Diagnosis of Pneumonia/Sepsis/Adult Respiratory Distress Syndrome (ARDS) | First 10 days of hospital stay
  Berlin classification for mild adult respiratory distress syndrome (previously ALI) and adult respiratory distress syndrome (ARDS). Centers for Disease Control and Prevention (CDC) definitions for pneumonia and sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Javier J Provencio, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No